CLINICAL TRIAL: NCT01809691
Title: A Phase III Randomized Trial Comparing Androgen Deprivation Therapy + TAK-700 With Androgen Deprivation Therapy + Bicalutamide in Patients With Newly Diagnosed Metastatic Sensitive Prostate Cancer
Brief Title: S1216, Phase III ADT+TAK-700 vs. ADT+Bicalutamide for Metastatic Prostate Cancer
Acronym: S1216
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1216; SWOG-S1216 (Other Grant/Funding Number: U10CA180888); NCI-2012-02876 (Other: NCI)
Record Dates: First submitted 2013-03-08; First posted 2013-03-13 (Estimated); Results first posted 2022-09-08 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; TAK-700; Bicalutamide; S1216; androgen therapy; Phase III
MeSH Terms: conditions — Prostatic Neoplasms | interventions — orteronel; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADT + TAK-700 (Experimental): LHRH agonist - given as approved for androgen deprivation at a dose necessary to maintain castrate levels and equivalent to 22.5 mg of Leuprolide IM every 3 months.
  TAK-700, 300 mg, PO, twice daily
  Interventions: Drug: TAK-700
- ADT + Bicalutamide (Active Comparator): LHRH agonist - given as approved for androgen deprivation at a dose necessary to maintain castrate levels and equivalent to 22.5 mg of Leuprolide IM every 3 months.
  Bicalutamide, 50 mg, PO, q daily
  Interventions: Drug: Bicalutamide

INTERVENTIONS:
Drug: TAK-700 — 300 mg, PO, twice daily
  Other Names: Orteronel
  Arms: ADT + TAK-700
Drug: Bicalutamide — 50 mg, PO, q daily
  Other Names: Casodex
  Arms: ADT + Bicalutamide

SUMMARY:
The purpose of this study is to compare overall survival in newly diagnosed metastatic prostate cancer patients randomly assigned to androgen deprivation therapy (ADT) + TAK-700 versus ADT + bicalutamide.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of metastatic prostate cancer.
* Serum testosterone within institutional limits of normal.
* PSA ≥ 2 ng/mL within 90 days prior to initiation of androgen deprivation. therapy (for early induction) or prior to registration (for late induction).
* DEXA scan within 2 years prior to registration.
* ECG within 42 days prior to registration and QTc interval ≤ 460 msec.
* LVEF within 42 days prior to registration and within institutional limits of normal.
* Adequate hepatic function as evidenced by bilirubin ≤ 2 x institutional upper limit of normal (ULN), SGOT (AST) and SGPT (ALT) ≤ 3 x institutional ULN, or ≤ 5 x institutional ULN if liver metastases are present.
* Adequate renal function as evidenced by calculated creatinine clearance ≥ 40 mL/min.
* Adequate hematologic function as evidenced by leukocytes ≥ 3,000/mcL, absolute neutrophil count (ANC) ≥ 1,500/mcL, hemoglobin ≥ 9 g/dL, and platelets ≥ 100,000/mcL.
* Zubrod performance status of 0 - 2. Zubrod performance status 3 will be allowed if from bone pain only.
* ≥ 18 years of age.
* Men of reproduction potential and those who are surgically sterilized (i.e., postvasectomy) must agree to practice effective barrier contraception or agree to abstain from intercourse while receiving treatment on this study and for at least 4 months after protocol treatment ends.

Exclusion Criteria:

* Known brain metastases.
* No more than 36 months of prior neoadjuvant and/or adjuvant hormonal therapy.
* ≥ 6 months since completion of androgen deprivation therapy.
* Prior or concurrent therapy with ketoconazole, aminoglutethimide or abiraterone acetate, or enzalutamide (MDV3100). Concurrent megestrol for hot flashes is allowed.
* Prior chemotherapy for treatment of metastatic prostate cancer. Prior chemotherapy in the neoadjuvant or adjuvant setting is allowed.
* ≥ 2 years since completion of chemotherapy in the neoadjuvant or adjuvant setting.
* Concurrent use of experimental therapy is not allowed.
* ≥ 30 days since prior medical castration for metastatic prostate cancer.
* If method of castration is a LHRH agonist, the patient must be willing to continue the use of LHRH and add bicalutamide or TAK-700 during protocol treatment.
* If the patient was on an antiandrogen (e.g. bicalutamide, flutamide), the patient must be willing to switch over to bicalutamide or TAK-700 (according to randomization).
* Prior bilateral orchiectomy.
* Concurrent use of LHRH antagonists (e.g. Degarelix)
* Grade III/IV cardiac disease (as defined by the NYHA Criteria), thromboembolic event, unstable angina pectoris, myocardial infarction within 6 months, or serious uncontrolled cardiac arrhythmia.
* Uncontrolled hypertension (defined as blood pressure > 160 mmHg systolic and > 90 mmHg diastolic at 2 separate measurements no more than 60 minutes apart during the Screening visit) despite appropriate medical therapy.
* Known human immunodeficiency virus (HIV)infection, active chronic hepatitis B or C, life-threatening illness unrelated to cancer, or any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with participation in this study.
* History of primary and secondary adrenal insufficiency.
* Hypersensitivity to TAK-700, to TAK-700 metabolites, to bicalutamide, or to LHRH agonists.
* Gastrointestinal (GI) disease or GI procedure that could interfere with the GI absorption or tolerance of TAK-700, including difficulty swallowing oral medications.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1313 (Actual)
Dates: Start 2013-03-08 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2025-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Agarwal, M.D., Principal Investigator — University of Utah
Locations (560):
- United States (560):
  - Veterans Administration Medical Center - Birmingham, Birmingham, Alabama
  - University of Arizona Cancer Center at Saint Joseph's, Phoenix, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Southern Arizona Veterans Affairs Health Center, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - Veteran's Administration Medical Center, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - City of Hope Corona, Corona, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fremont, Fremont, California
  - University Oncology Associates, Fresno, California
  - Kaiser Permanente, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Loma Linda Healthcare System, Loma Linda, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mather Veteran Affairs Medical Center, Mather, California
  - Mercy UC Davis Cancer Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - PCR Oncology, Pismo Beach, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Northbay Cancer Center, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Greenwich Hospital, Greenwich, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center -Washington DC, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Presence Saint Joseph Hospital-Chicago, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Hines Veterans Administration Hospital, Hines, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health Bloomington, Bloomington, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Porter Memorial Hospital, Valparaiso, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Iowa City VA Healthcare System, Iowa City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Heartland Cancer Center, Great Bend, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Topeka VA Hospital, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Montgomery General Hospital-Olney, Olney, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Steward Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Dana Farber Community Cancer Care-Quincy, Quincy, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton Health Center, Canton, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Botsford General Hospital, Farmington, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis Veterans Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center - Saint Peters, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Barnes-Jewish West County Hospital, Creve Coeur, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - The University of Kansas Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Lovelace Medical Center-Downtown, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Veteran Affairs New York Harbor Healthcare System-Brooklyn Campus, Brooklyn, New York
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Carolinas HealthCare System NorthEast, Concord, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Carolinas HealthCare System Union, Monroe, North Carolina
  - Carolinas HealthCare System Cleveland, Shelby, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Wright-Patterson Medical Center, Wpafb, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Portland Veterans Administration Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates-Roper, Charleston, South Carolina
  - Charleston Hematology Oncology Associates PA-St. Francis, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - MD Anderson Regional Care Center-Katy, Houston, Texas
  - MD Anderson Regional Care Center-Bay Area, Nassau Bay, Texas
  - MD Anderson Regional Care Center-Sugar Land, Sugar Land, Texas
  - MD Anderson Regional Care Center-The Woodlands, The Woodlands, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Memorial Hospital Of Martinsville, Martinsville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology Associates PC, Winchester, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
https://swog.org/Visitors/Download/Policies/Policy43.pdf

REFERENCES:
- [Derived] Gebrael G, Jo Y, Swami U, Plets M, Hage Chehade C, Narang A, Gupta S, Myint ZW, Sayegh N, Tangen CM, Hussain M, Dorff T, Lara PN Jr, Lerner SP, Thompson I, Agarwal N. Bone Pain and Survival Among Patients With Metastatic, Hormone-Sensitive Prostate Cancer: A Secondary Analysis of the SWOG-1216 Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2419966. doi: 10.1001/jamanetworkopen.2024.19966. PMID 38980676
- [Derived] Lara PN Jr, Mayerson E, Gertz E, Tangen C, Goldkorn A, van Loan M, Hussain M, Gupta S, Zhang J, Parikh M, Twardowski P, Quinn DI, LeBlanc M, Thompson I, Agarwal N. Markers of bone metabolism and overall survival in men with bone-metastatic hormone sensitive prostate cancer (HSPC): A subset analysis of SWOG S1216, a phase III trial of androgen deprivation with or without orteronel. Prostate Cancer Prostatic Dis. 2024 Sep;27(3):566-570. doi: 10.1038/s41391-024-00813-3. Epub 2024 Feb 29. PMID 38424319
- [Derived] Sayegh N, Swami U, Jo Y, Gebrael G, Haaland B, Gupta S, Plets M, Hussain MHA, Quinn DI, Lara PN Jr, Thompson IM Jr, Agarwal N. Race and Treatment Outcomes in Patients With Metastatic Castration-Sensitive Prostate Cancer: A Secondary Analysis of the SWOG 1216 Phase 3 Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2326546. doi: 10.1001/jamanetworkopen.2023.26546. PMID 37526936
- [Derived] Agarwal N, Tangen CM, Hussain MHA, Gupta S, Plets M, Lara PN, Harzstark AL, Twardowski PW, Paller CJ, Zylla D, Zibelman MR, Levine E, Roth BJ, Goldkorn A, Vaena DA, Kohli M, Crispino T, Vogelzang NJ, Thompson IM Jr, Quinn DI. Orteronel for Metastatic Hormone-Sensitive Prostate Cancer: A Multicenter, Randomized, Open-Label Phase III Trial (SWOG-1216). J Clin Oncol. 2022 Oct 1;40(28):3301-3309. doi: 10.1200/JCO.21.02517. Epub 2022 Apr 21. PMID 35446628
- See also: Related Info — https://nctn-data-archive.nci.nih.gov/
- Available data/document: Individual Participant Data Set — https://nctn-data-archive.nci.nih.gov/ — Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1,313 participants were enrolled and randomly assigned. 32 participants were deemed ineligible and 2 withdrew consent before starting treatment. Therefore, 1,279 were deemed eligible and analyzable for the primary analysis.
Groups:
- LHRHa + TAK-700: Experimental: ADT + TAK-700 LHRH agonist - given as approved for androgen deprivation at a dose necessary to maintain castrate levels and equivalent to 22.5 mg of Leuprolide IM every 3 months.
  TAK-700, 300 mg, PO, twice daily
- LHRHa + Bicalutamide: Active Comparator: ADT + Bicalutamide LHRH agonist - given as approved for androgen deprivation at a dose necessary to maintain castrate levels and equivalent to 22.5 mg of Leuprolide IM every 3 months.
  Bicalutamide, 50 mg, PO, q daily
Period: Overall Study
Arm/Group | LHRHa + TAK-700 | LHRHa + Bicalutamide
Started | 638 | 641
Completed | 0 | 0
Not Completed | 638 | 641
Not completed — Currently on Treatment | 192 | 100
Not completed — No Protocol Treatment | 10 | 11
Not completed — Adverse Event | 80 | 21
Not completed — Disease Progression | 226 | 372
Not completed — Death | 26 | 13
Not completed — Participant Refusal | 70 | 72
Not completed — Other, Not Specified | 34 | 52

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LHRHa + TAK-700 | LHRHa + Bicalutamide | Total
Number analyzed (Participants) | 638 | 641 | 1279
Age, Continuous [Median (Full Range); unit: years] | 67.6 [46.1 to 90.0] | 68.1 [19.4 to 92.3] | 67.8 [19.4 to 92.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 638 | 641 | 1279
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 539 | 538 | 1077
  Black | 64 | 71 | 135
  Others | 35 | 32 | 67
Zubrod Performance Status Score [Count of Participants; unit: Participants] — Zubrod performance status scores range from 0 to 3, with higher scores reflecting greater disability.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  3. Capable of limited self-care, confined to bed or chair more than 50% of waking hours.
  Participants
    0 | 416 | 442 | 858
    1 | 197 | 175 | 372
    2 | 21 | 21 | 42
    3 | 3 | 2 | 5
    Missing | 1 | 1 | 2
Gleason Score at Initial Diagnosis [Count of Participants; unit: Participants] — Gleason scores can range from 2 to 10, but most often range from 6 to 10. A higher Gleason score indicates a more well-differentiated, aggressive tumor.
  Participants
    < 7 | 46 | 39 | 85
    7 | 165 | 168 | 333
    8 | 123 | 118 | 241
    9-10 | 249 | 264 | 513
    Missing | 55 | 52 | 107
Median PSA Level [Median (Full Range); unit: ng/mL] | 27.2 [2.0 to 6710.0] | 31.8 [2.0 to 6651.2] | 29.7 [2.0 to 6710.0]
Bone Pain [Count of Participants; unit: Participants]
  Yes | 158 | 143 | 301
  No | 480 | 498 | 978
Bone Metastases [Count of Participants; unit: Participants]
  Yes | 470 | 482 | 952
  No | 168 | 159 | 327
Liver Metastases [Count of Participants; unit: Participants]
  Yes | 16 | 14 | 30
  No | 622 | 627 | 1249
Other Visceral Metastases [Count of Participants; unit: Participants]
  Yes | 82 | 72 | 154
  No | 556 | 569 | 1125
Disease Severity [Count of Participants; unit: Participants]
  Minimal | 328 | 328 | 656
  Extensive | 310 | 313 | 623
Preregistration LHRH Suppression [Count of Participants; unit: Participants]
  Yes | 330 | 331 | 661
  No | 308 | 310 | 618
Bisphosphonate Use at Study Entry [Count of Participants; unit: Participants]
  Yes | 39 | 35 | 74
  No | 599 | 606 | 1205
Prior Radical Prostatectomy [Count of Participants; unit: Participants]
  Yes | 167 | 148 | 315
  No | 471 | 493 | 964
Prior Bilateral Orchiectomy [Count of Participants; unit: Participants]
  Yes | 4 | 3 | 7
  No | 634 | 638 | 1272

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from random assignment to the date of death from any cause
Time Frame: Duration of treatment and follow-up until death or 9 years after study start
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LHRHa + TAK-700 | LHRHa + Bicalutamide
Number analyzed (Participants) | 638 | 641
months | 81.1 [68.0 to NA] — Not enough event data to estimate the upper bound of the 95% CI for median OS for the TAK700 arm. | 70.2 [64.6 to 79.5]
Statistical Analysis 1: Comparison: LHRHa + TAK-700 vs LHRHa + Bicalutamide; Test type: Superiority; p = .080, Regression, Cox; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.72 to 1.02]

2. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS) is defined as the time from random assignment to first documentation of PSA progression, radiologic progression, clinical progression, or death, whichever occurred first.
  PSA progression is defined as a ≥25% increase AND and absolute increase of at last 2 ng/mL from the nadir PSA (or from baseline PSA if there was no drop in PSA after starting treatment).
  Radiologic progression is defined as two or more new lesions on radionuclide bone scans.
  Clinical progression is defined using the Response Evaluation Criteria in Solid Tumors (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Duration of treatment and follow-up until death or 9 years after study start
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LHRHa + TAK-700 | LHRHa + Bicalutamide
Number analyzed (Participants) | 638 | 641
months | 47.6 [42.2 to 54.2] | 23.0 [19.3 to 26.3]
Statistical Analysis 1: Comparison: LHRHa + TAK-700 vs LHRHa + Bicalutamide; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.51 to 0.67]

3. Secondary Outcome: PSA Response Rates
Description: Prostate-specific antigen (PSA) response rates were divided into complete response (CR: PSA < 0.2 ng/mL), partial response (PR: PSA between 0.2 and 4.0 ng/mL), and no response (NR: PSA > 4.0 ng/mL) at a 7-month landmark after random assignment.
Time Frame: 7 months after randomization
Measure: Number; unit: percentage of participants
Arm/Group | LHRHa + TAK-700 | LHRHa + Bicalutamide
Number analyzed (Participants) | 638 | 641
percentage of participants
  Complete Response | 58 | 44
  Partial Response | 22 | 31
  No Response | 19 | 25

4. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported. Adverse events are graded using the Common Terminology Criteria for Adverse Events (CTCAE v4.0) where grade refers to the severity of the AE.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care.
  Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE.
Time Frame: Duration of treatment and follow-up until death or 9 years after study start
Population: Eligible participants who received at least one dose of protocol treatment
Measure: Number; unit: Participants
Arm/Group | LHRHa + TAK-700 | LHRHa + Bicalutamide
Number analyzed (Participants) | 627 | 629
Participants
  Abdominal pain | 4 | 0
  Acute coronary syndrome | 1 | 1
  Acute kidney injury | 0 | 2
  Adrenal insufficiency | 2 | 0
  Adult respiratory distress syndrome | 1 | 0
  Agitation | 0 | 1
  Alanine aminotransferase increased | 10 | 2
  Alkaline phosphatase increased | 9 | 3
  Allergic reaction | 2 | 0
  Anaphylaxis | 1 | 0
  Anemia | 1 | 2
  Anorexia | 4 | 1
  Anxiety | 1 | 2
  Arthralgia | 5 | 2
  Arthritis | 1 | 0
  Aspartate aminotransferase increased | 7 | 3
  Atrial fibrillation | 8 | 0
  Back pain | 1 | 0
  Blood bilirubin increased | 4 | 1
  Bone pain | 0 | 3
  Cardiac arrest | 0 | 1
  Cardiac disorders - Other, specify | 1 | 0
  Cardiac troponin I increased | 1 | 0
  Chest pain - cardiac | 4 | 0
  Colitis | 2 | 0
  Concentration impairment | 1 | 0
  Confusion | 1 | 1
  Constipation | 2 | 0
  Creatinine increased | 1 | 1
  Death NOS | 1 | 0
  Dehydration | 2 | 1
  Depression | 7 | 2
  Diarrhea | 10 | 2
  Dizziness | 3 | 1
  Dysphagia | 1 | 0
  Dyspnea | 9 | 1
  Edema limbs | 4 | 0
  Ejection fraction decreased | 1 | 0
  Encephalopathy | 1 | 1
  Erectile dysfunction | 4 | 4
  Esophagitis | 1 | 0
  Fall | 2 | 0
  Fatigue | 34 | 11
  Fever | 1 | 0
  Flank pain | 1 | 0
  Flu like symptoms | 1 | 0
  GGT increased | 1 | 0
  Gastric hemorrhage | 1 | 0
  Gastric ulcer | 1 | 0
  General disorders and admin site conditions - Other | 0 | 1
  Generalized muscle weakness | 4 | 1
  Gynecomastia | 1 | 0
  Headache | 3 | 1
  Heart failure | 6 | 2
  Hematuria | 1 | 2
  Hepatobiliary disorders - Other, specify | 1 | 0
  Hip fracture | 3 | 0
  Hoarseness | 0 | 1
  Hot flashes | 5 | 5
  Hyperglycemia | 11 | 6
  Hyperkalemia | 2 | 0
  Hypertension | 127 | 28
  Hypertriglyceridemia | 1 | 3
  Hyperuricemia | 1 | 0
  Hypokalemia | 20 | 1
  Hyponatremia | 5 | 1
  Hypophosphatemia | 0 | 1
  Hypotension | 2 | 1
  Hypoxia | 2 | 0
  Infections and infestations - Other, specify | 2 | 0
  Insomnia | 2 | 1
  Investigations - Other, specify | 1 | 0
  Joint infection | 1 | 0
  Laryngeal edema | 1 | 0
  Left ventricular systolic dysfunction | 2 | 0
  Leukocytosis | 1 | 0
  Lipase increased | 9 | 0
  Lung infection | 5 | 0
  Lymphocyte count decreased | 3 | 0
  Mucositis oral | 1 | 0
  Multi-organ failure | 0 | 1
  Muscle weakness lower limb | 0 | 2
  Musculoskeletal and connective tiss disorder - Other | 3 | 0
  Myalgia | 1 | 0
  Myocardial infarction | 5 | 0
  Nausea | 5 | 0
  Neutrophil count decreased | 1 | 1
  Obesity | 0 | 2
  Osteoporosis | 1 | 1
  Otitis media | 1 | 0
  Pain | 3 | 1
  Pancreatitis | 7 | 0
  Peripheral sensory neuropathy | 1 | 0
  Platelet count decreased | 0 | 1
  Pneumonitis | 1 | 0
  Pruritus | 1 | 0
  Pulmonary edema | 1 | 0
  Pulmonary hypertension | 1 | 0
  Renal calculi | 0 | 2
  Resp, thoracic and mediastinal disorders - Other | 2 | 0
  Serum amylase increased | 2 | 0
  Skin and subcutaneous tissue disorders - Other | 1 | 0
  Spinal fracture | 0 | 1
  Stroke | 2 | 1
  Supraventricular tachycardia | 1 | 0
  Syncope | 4 | 3
  Thromboembolic event | 6 | 0
  Thrombotic thrombocytopenic purpura | 1 | 0
  Urinary tract infection | 4 | 1
  Urostomy stenosis | 0 | 1
  Ventricular fibrillation | 1 | 0
  Ventricular tachycardia | 1 | 0
  Vomiting | 4 | 0
  Weight gain | 3 | 2
  Weight loss | 4 | 1

5. Secondary Outcome: Long-term Survival
Description: Long-term survival is defined as the time from random assignment to the date of death from any cause
Time Frame: After 10 years of follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow-up until death or 9 years after study start
Description: 1,256 eligible participants who received protocol treatment were evaluable for AEs: 627 on the LHRHa + TAK-700 arm and 629 on the LHRHa + Bicalutamide arm. Adverse Events (AEs) and Serious Adverse Events (SAEs) are reported by CTCAE Version 4.0. All 1,279 participants who started the study, 638 on the LHRHa + TAK-700 arm and 641 on the LHRHa + Bicalutamide arm, were evaluated for All-Cause Mortality.
Arm/Group | LHRHa + TAK-700 | LHRHa + Bicalutamide
All-Cause Mortality (participants affected / at risk) | 251/638 | 274/641
Serious Adverse Events (participants affected / at risk) | 235/627 | 15/629
Other Adverse Events (participants affected / at risk) | 615/627 | 609/629
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LHRHa + TAK-700 (N=627) | LHRHa + Bicalutamide (N=629)
Anemia (Blood and lymphatic system disorders) | 6 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 3 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 18 | 0
Cardiac arrest (Cardiac disorders) | 6 | 2
Cardiac disorders-Other (Cardiac disorders) | 5 | 0
Chest pain - cardiac (Cardiac disorders) | 16 | 0
Heart failure (Cardiac disorders) | 12 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 10 | 0
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Blurred vision (Eye disorders) | 3 | 0
Retinal detachment (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 16 | 0
Colitis (Gastrointestinal disorders) | 4 | 0
Colonic hemorrhage (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 10 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 2 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 4 | 0
Ileal obstruction (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 10 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 8 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 10 | 0
Chills (General disorders) | 1 | 0
Death NOS (General disorders) | 5 | 2
Edema face (General disorders) | 1 | 0
Edema limbs (General disorders) | 4 | 0
Fatigue (General disorders) | 10 | 0
Fever (General disorders) | 10 | 0
Flu like symptoms (General disorders) | 3 | 0
Gait disturbance (General disorders) | 2 | 0
General disorders and admin site conditions - Other (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 6 | 0
Pain (General disorders) | 1 | 0
Sudden death NOS (General disorders) | 5 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 0
Anaphylaxis (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Anorectal infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Bone infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Infections and infestations-Other (Infections and infestations) | 10 | 1
Lung infection (Infections and infestations) | 24 | 0
Otitis media (Infections and infestations) | 1 | 0
Prostate infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 7 | 0
Skin infection (Infections and infestations) | 4 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 14 | 0
Wound infection (Infections and infestations) | 5 | 0
Aortic injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 9 | 0
Fracture (Injury, poisoning and procedural complications) | 5 | 0
Hip fracture (Injury, poisoning and procedural complications) | 7 | 0
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 2 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 7 | 0
Alkaline phosphatase increased (Investigations) | 5 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 0
Blood bilirubin increased (Investigations) | 6 | 0
Cardiac troponin I increased (Investigations) | 2 | 0
Creatinine increased (Investigations) | 2 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 | 0
Investigations-Other (Investigations) | 2 | 0
Lipase increased (Investigations) | 11 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 0
Serum amylase increased (Investigations) | 4 | 0
Weight loss (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 8 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 12 | 0
Hyponatremia (Metabolism and nutrition disorders) | 5 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 5 | 0
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Ataxia (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 8 | 0
Encephalopathy (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 4 | 0
Intracranial hemorrhage (Nervous system disorders) | 3 | 0
Lethargy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 10 | 1
Syncope (Nervous system disorders) | 13 | 0
Transient ischemic attacks (Nervous system disorders) | 2 | 0
Vasovagal reaction (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 4 | 1
Delirium (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 4 | 0
Hallucinations (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 9 | 0
Cystitis noninfective (Renal and urinary disorders) | 2 | 0
Hematuria (Renal and urinary disorders) | 8 | 0
Renal and urinary disorders-Other (Renal and urinary disorders) | 3 | 0
Renal calculi (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 4 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 23 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Surgical and medical procedures-Other (Surgical and medical procedures) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 44 | 0
Hypotension (Vascular disorders) | 7 | 0
Thromboembolic event (Vascular disorders) | 20 | 0
Vascular disorders-Other (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LHRHa + TAK-700 (N=627) | LHRHa + Bicalutamide (N=629)
Anemia (Blood and lymphatic system disorders) | 340 | 271
Sinus tachycardia (Cardiac disorders) | 36 | 15
Abdominal pain (Gastrointestinal disorders) | 88 | 50
Constipation (Gastrointestinal disorders) | 228 | 133
Diarrhea (Gastrointestinal disorders) | 181 | 90
Dry mouth (Gastrointestinal disorders) | 46 | 16
Dyspepsia (Gastrointestinal disorders) | 36 | 14
Flatulence (Gastrointestinal disorders) | 41 | 20
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 38 | 17
Nausea (Gastrointestinal disorders) | 214 | 86
Vomiting (Gastrointestinal disorders) | 120 | 47
Chills (General disorders) | 33 | 19
Edema limbs (General disorders) | 150 | 110
Fatigue (General disorders) | 445 | 346
Flu like symptoms (General disorders) | 41 | 34
General disorders and admin site conditions - Other (General disorders) | 61 | 47
Non-cardiac chest pain (General disorders) | 47 | 25
Pain (General disorders) | 208 | 156
Infections and infestations-Other (Infections and infestations) | 57 | 26
Upper respiratory infection (Infections and infestations) | 45 | 29
Urinary tract infection (Infections and infestations) | 48 | 26
Fall (Injury, poisoning and procedural complications) | 62 | 34
Alanine aminotransferase increased (Investigations) | 179 | 85
Alkaline phosphatase increased (Investigations) | 135 | 107
Aspartate aminotransferase increased (Investigations) | 182 | 86
Blood bilirubin increased (Investigations) | 40 | 36
Cholesterol high (Investigations) | 51 | 52
Creatinine increased (Investigations) | 151 | 99
Investigations-Other (Investigations) | 49 | 21
Lymphocyte count decreased (Investigations) | 128 | 52
Neutrophil count decreased (Investigations) | 38 | 32
Platelet count decreased (Investigations) | 95 | 60
Weight gain (Investigations) | 66 | 103
Weight loss (Investigations) | 130 | 38
White blood cell decreased (Investigations) | 90 | 55
Anorexia (Metabolism and nutrition disorders) | 134 | 60
Hypercalcemia (Metabolism and nutrition disorders) | 53 | 54
Hyperglycemia (Metabolism and nutrition disorders) | 244 | 172
Hyperkalemia (Metabolism and nutrition disorders) | 73 | 36
Hypernatremia (Metabolism and nutrition disorders) | 62 | 30
Hypertriglyceridemia (Metabolism and nutrition disorders) | 85 | 58
Hypoalbuminemia (Metabolism and nutrition disorders) | 58 | 25
Hypocalcemia (Metabolism and nutrition disorders) | 63 | 32
Hypokalemia (Metabolism and nutrition disorders) | 130 | 37
Hyponatremia (Metabolism and nutrition disorders) | 87 | 59
Arthralgia (Musculoskeletal and connective tissue disorders) | 157 | 101
Arthritis (Musculoskeletal and connective tissue disorders) | 53 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 213 | 194
Bone pain (Musculoskeletal and connective tissue disorders) | 66 | 74
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 103 | 55
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 85 | 62
Myalgia (Musculoskeletal and connective tissue disorders) | 101 | 63
Neck pain (Musculoskeletal and connective tissue disorders) | 47 | 36
Osteoporosis (Musculoskeletal and connective tissue disorders) | 51 | 28
Pain in extremity (Musculoskeletal and connective tissue disorders) | 220 | 147
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 | 19
Dizziness (Nervous system disorders) | 152 | 99
Dysgeusia (Nervous system disorders) | 51 | 16
Headache (Nervous system disorders) | 190 | 84
Memory impairment (Nervous system disorders) | 43 | 27
Peripheral sensory neuropathy (Nervous system disorders) | 103 | 70
Anxiety (Psychiatric disorders) | 90 | 51
Depression (Psychiatric disorders) | 118 | 80
Insomnia (Psychiatric disorders) | 169 | 96
Libido decreased (Psychiatric disorders) | 33 | 40
Hematuria (Renal and urinary disorders) | 58 | 38
Renal and urinary disorders-Other (Renal and urinary disorders) | 58 | 37
Urinary frequency (Renal and urinary disorders) | 155 | 114
Urinary incontinence (Renal and urinary disorders) | 69 | 53
Urinary retention (Renal and urinary disorders) | 40 | 22
Erectile dysfunction (Reproductive system and breast disorders) | 62 | 70
Gynecomastia (Reproductive system and breast disorders) | 43 | 72
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 33 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 152 | 85
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 147 | 90
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 51 | 29
Alopecia (Skin and subcutaneous tissue disorders) | 35 | 31
Dry skin (Skin and subcutaneous tissue disorders) | 55 | 27
Pruritus (Skin and subcutaneous tissue disorders) | 55 | 19
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 77 | 38
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 68 | 44
Hot flashes (Vascular disorders) | 448 | 453
Hypertension (Vascular disorders) | 364 | 222
Hypotension (Vascular disorders) | 35 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT01809691/Prot_SAP_ICF_000.pdf